CLINICAL TRIAL: NCT05518864
Title: GAG-therapy Efficacy Trial Solution for Bladder Pain Syndrome/ Interstitial Cystitis
Brief Title: GAG-therapy Efficacy Trial Solution for Bladder Pain Syndrome/ Interstitial Cystitis (GETSBI Study)
Acronym: GETSBI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); IQ Healthcare (Unknown); Radboud Technology Ceter (Unknown); Zorginstituut Nederland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 110130
Record Dates: First submitted 2020-12-21; First posted 2022-08-29 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-02

CONDITIONS: Bladder Pain Syndrome
Keywords: Bladder Pain Syndrome; GAG therapy; Hunner lesion; RCT; N-of-1 trial
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Study start as a normal double blinded RCT, but continues with an aggregated N-of-1 (multi-crossover) type trial
Who Masked: Participant, Care Provider
Masking Description: double blinded by care provider (person giving the treatment) and the participant (blinded syringes en placebo product)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo - Intervention - Intervention (Experimental): Treatment period 1: placebo for 1x/week for 6 weeks, followed by two treatment periods of 6 weeks receiving GAG-therapy (Ialuril) 1x/week.
  Finally this arm continues with unblinded GAG-therapy (Ialuril) instillations 1x/month for 6 instillations.
  Interventions: Device: IALURIL Prefill
- Intervention - Placebo - Intervention (Experimental): Treatment period 1: GAG-therapy (Ialuril) for 1x/week for 6 weeks, followed by treatment period 2: Placebo for 1x/week for 6 weeks and afterwards treatment period 3: GAG-therapy (Ialuril) for 1/x week for 6 weeks.
  Finally, this arm continues with unblinded GAG-therapy (Ialuril) instillations 1x/month for 6 instillations.
  Interventions: Device: IALURIL Prefill
- Intervention - Intervention - Placebo (Experimental): Treatment period 1: GAG-therapy (Ialuril) for 1x/week for 6 weeks, followed by treatment period 2: GAG-therapy (Ialuril) for 1x/week for 6 weeks and afterwards treatment period 3: placebo for 1/x week for 6 weeks.
  Finally, this arm continues with unblinded GAG-therapy (Ialuril) instillations 1x/month for 6 instillations.
  Interventions: Device: IALURIL Prefill

INTERVENTIONS:
Device: IALURIL Prefill — GAG therapy (bladder instillations with glycosaminoglycans)

SUMMARY:
Rationale:

Efficacy study (RCT) for glycosaminoglycan(GAG)-therapy for the indication bladder pain syndrome / interstitial cystitis with Hunner lesion subtype (BPS-IC H+). reason for this study is a current lack of evidence regarding its efficacy and cost-effectiveness.

Main objective is to determine short and long term efficacy of GAG therapy (bladder instillations) for people with BPS-IC H+ as compared to placebo treatment on dominant symptoms such as pain and Quality of Life (QOL)

DETAILED DESCRIPTION:
Rationale:

Reimbursement in the Netherlands for GAG-therapy for bladder pain syndrome / interstitial cystitis patients with Hunner lesion subtype (BPS-IC H+) is under debate, as evidence regarding its efficacy and cost-effectiveness is lacking.

Objective:

Main objective is to determine short and long term efficacy of GAG therapy (bladder instillations) for people with BPS-IC H+ as compared to placebo treatment on dominant symptoms such as pain. Secondary objectives are to determine the 1) cost-effectiveness of GAG therapy, 2) effectiveness of GAG therapy on quality of life and bladder inflammation evaluated by urethrocystoscopy

Study design:

Multi-design study. Study is powered and set-up as double-blinded randomized intervention study and is extended with a double-blinded aggregated N-of-1 trial. As requested by the Zorginstituut Netherlands, the study will be further extended with a prospective, non-blinded intervention study to evaluate long term follow up with a low frequency therapy dose.

Study population:

People with symptomatic BPS-IC H+ (> 18 yrs old). A total of 80 patients will be included for the main study.

Intervention :

GAG bladder instillations (hyaluronic acid + chondroitin sulfate; Ialuril) 50ml administered with a catheter. Placebo will be Hypromellose 50ml administered with a catheter. Patients will receive instillations (Ialuril / placebo with ratio 2:1) in 3 periods of 6 wks with frequency of 1 instillation/wk. With wash-out periods 4 wks. After 3 periods of treatment / placebo (wk 30), blinding will cease and continue unblinded where all subjects will receive maintenance therapy Ialuril for 1x/4wk until 54 weeks (endpoint).

Main study parameters/endpoints:

Primary outcome parameter: change from baseline in maximum bladder pain (visual analogue scale (VAS) pain score (3d average and maximal pain score).

Secondary outcome parameters:

* Change from baseline in VAS score (0-10) on self-reported secondary symptoms
* Change from baseline from self-reported Global Assessment of Improvement (Likert scale)
* Change from baseline from O'Leary-Sant IC Symptom Index & Problem Index questionnaire
* Change from baseline in urethrocystoscopic evaluation of bladder mucosa (inflammation, active Hunner lesions) (clinician assessed estimated % of inflammation & degree of inflammation)
* Change from baseline in Quality of Life using ED-5D 5L questionnaire (Dutch)
* Cost effectiveness analyses using iMCQ and iPCQ questionnaires
* Changes in Patient Reported Outcome questionnaire (incl. urinary frequency)
* Adverse events using Clavien-Dindo system

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Benefits patients and group relatedness. All participants are capacitated adults and will receive a similar amount of intervention and placebo treatments. Treatment corresponds to the Dutch NVU guideline BPS. Therapy will be reimbursed for patients. During 54wks, patients will have a 6 week period where placebo is given. Due to the study design, patients can obtain a personal (individual) study efficacy result if therapy was successful in him/her.

Therapy and placebo: risks and burden This study will be submitted as low-intervention trial. GAG therapy (instillations) has been used for >25 yrs in clinical practice to treat BPS-IC. GAG-therapies are registered as medical devices. The therapy is instilled into the bladder using a catheter (by nurse / patient). Catherization has a small increased risk for developing an urine tract infection (1.9%) [Herr 2015], urethral discomfort and in rare cases urethral trauma.

The placebo compound Hypromellose 0.3% is used as moisturizing drops to treat dry eyes. It is inert (non-irritating and hypo-allergenic). Very rare (< 0.01%) side effects are reported in the Dutch 'Farmacologisch Kompas'. They report local side effects of sensitivity (burning, itch, tears e.d.). Blurry vision. and very rare systemic effects as rash, itch.Because of these reported side effects at inclusion the (over)sensitivity is checked by one drop in an eye, taking into account the possible blurry vision afterwards.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 yrs or older) with symptomatic BPS with established Hunner lesions objectified with urethrocystoscopy in the 3 months prior to inclusion.
2. A VAS pain score (maximum pain during the last 3 days; scale 0-10) of at least 4.

Exclusion Criteria:

1. pain, discomfort in pelvic region of inflammatory bladder conditions due to any cause other than BPS with Hunner lesions, with the exception of irritable bowel syndrome (IBS) and hypertonic pelvic floor or urine tract infections (UTI; <3 UTI's / year). This is noted by ESSIC as a confusable disease [van de Merwe 2007, contains an elaborate table for this].
2. had a urine tract infection in the previous 6 weeks.
3. received bladder instillations for BPS in the previous 3 months;
4. received intradetrusor Botulinum toxin (BOTOX) injections within the previous 12 months.
5. received transurethral coagulation/ablation therapy of Hunner lesions within the last 12 months, with the exception of patients who have objectified Hunner lesion recurrence(s) on cystoscopy after coagulation/ablation therapy after at least 3 months' post-intervention.
6. started a new treatment for (chronic) pain (pharmacotherapy) or urine tract infection in the last month.
7. Unable (also legal) to give informed consent.
8. Allergic to Hypromellose (tested in one eye)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-10-21 (Estimated); Study Completion 2024-10-21 (Estimated)

PRIMARY OUTCOMES:
Change in maximum bladder pain | Fase 1: Week 1,2,5,7,8,12,15,17,18,22,25,27,28,29 Fase 2:week 32, 36, 40, 44, 48, 54
  VAS pain score (0-10; 0= no pain, 10=worst pain)

SECONDARY OUTCOMES:
Change in average bladder pain | Fase 1: Week 1,2,5,7,8,12,15,17,18,22,25,27,28,29 Fase 2:week 32, 36, 40, 44, 48, 54
  VAS pain score (0-10; 0= no pain, 10=worst pain)
7-point Global Response Assessment (GRA) scale | Fase 1: Week 1,2,5,7,8,12,15,17,18,22,25,27,28,29 Fase 2:week 32, 36, 40, 44, 48, 54
  The GRA is a 7-point descriptive scale, scores of 1-3 indicate worsening of symptoms, and 5-7 indicate and improvement in symptoms
Change in patient assessed most dominant symptom | Fase 1: Week 1,2,5,7,8,12,15,17,18,22,25,27,28,29 Fase 2:week 32, 36, 40, 44, 48, 54
  VAS score (0-10; 0= no burden, 10=high burden)
Voiding urgency | Fase 1: Week 1,2,5,7,8,12,15,17,18,22,25,27,28,29 Fase 2:week 32, 36, 40, 44, 48, 54
  as single item from the validated Genito-Urinary Pain Index questionnaire (5 point Likert scale)
Voiding frequency | Fase 1: Week 1,2,5,7,8,12,15,17,18,22,25,27,28,29 Fase 2:week 32, 36, 40, 44, 48, 54
  as single item from the validated Genito-Urinary Pain Index questionnaire (5 point Likert scale)
O'leary Sant interstitial cystitis symptom index/problem index (ICSI/ICPI) | week 1, 6, 18, 28, 29, 40, 48
  Validated BPS-IC related symptom questionaire
Patient Reported Outcome Measurement (PROM) short and extended | week 1, 8, 18, 28, 29, 40, 48
  Improvement (0-100%), continue treatment, reccommend to family, including Adverse Events and start/stop other treatment for BPS/IC
Voiding diary | at baseline
  2x24h
Quality of Life questionnaire | week 1, 6, 18, 28, 29, 40, 48
  Outcome of ED-5D 5L QoL questionnaire
Urine sediment | week 1, 6, 18, 28, 29, 40, 48
  Screening for bacterial urinary tract infection
Cost effectiveness | week 1, 8, 18, 28
  iMCQ and iPCQ questionaires
Cystoscopic evaluation | week 8 and week 28
  Likert scale inflammation (1-5)

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Radboud Unviversity Nijmegen Medical Centre, Nijmegen, Gelderland
  - Rijnstate, Arnhem
  - Andros Clinics, Baarn
  - Slingeland, Doetinchem
  - Catharina ziekenhuis, Eindhoven
  - Alrijne ziekenhuis, Leiden
  - MUMC+, Maastricht
  - Isala klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No
only anonymous patient data will be shared

REFERENCES:
- [Derived] van Ginkel C, Groenewoud JMM, Hoogeboom TJ, Heesakkers J, Martens F, Janssen D. Carry-over effects in GAG therapy efficacy trial solution for bladder pain syndrome/interstitial cystitis (GETSBI study): an interim analysis. BMJ Open. 2025 Jun 5;15(6):e092757. doi: 10.1136/bmjopen-2024-092757. PMID 40473282
- [Derived] van Ginkel C, Baars C, Heesakkers J, Martens F, Janssen D. Study protocol of a multicentre double-blind RCT, comparing a traditional RCT with an aggregated N-of-1 trial: GAG therapy Efficacy Trial Solution for Bladder pain syndrome/Interstitial cystitis (GETSBI study). BMJ Open. 2023 Apr 12;13(4):e068546. doi: 10.1136/bmjopen-2022-068546. PMID 37045569